CLINICAL TRIAL: NCT00531219
Title: Natural Orifice Translumenal Endoscopic Surgery (NOTES): Laparoscopic Assisted Transgastric Appendectomy and Cholecystectomy
Brief Title: Minimally Invasive Surgery: Using Natural Orifice Translumenal Endoscopic Surgery (NOTES)
Acronym: NOTES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Santiago Horgan, Professor of Surgery, University of California, San Diego
Other Study IDs: 071114, 140016
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Appendicitis; Cholelithiasis
Keywords: appendicitis; cholelithiasis; gallstones
MeSH Terms: conditions — Appendicitis; Cholelithiasis; Gallstones

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Group #1 NOTES Appendectomy - Transgastric approach
  Interventions: Procedure: Transgastric Appendectomy
- 2: Group #2 NOTES Cholecystectomy - Transgastric approach
  Interventions: Procedure: Transgastric Cholecystectomy

INTERVENTIONS:
Procedure: Transgastric Appendectomy — The appendix will be removed through an incision in the stomach and pulled out through the mouth
  Groups: 1
Procedure: Transgastric Cholecystectomy — The gallbladder will be removed through an incision in the stomach and pulled out through the mouth.
  Groups: 2

SUMMARY:
This is an observational study of pain and outcomes from patients undergoing transgastric NOTES removal of their appendix or gallbladder. Subjects who elect to have a transgastric NOTES removal of their appendix or gallbladder and agree to be in this study (through signature on the informed consent form) will be followed per standard of care, with additional follow-up for data collection including the following:

* Subjects will complete a 7 day pain/temperature log after surgery
* Subjects will receive a phone call at 6 months and at 1 year after surgery to capture data related to safety, adverse events, hospitalizations and patient satisfaction

Additional data related to pain and outcomes will be collected at baseline/screening and at follow-up as necessary.

ELIGIBILITY:
Inclusion criteria for the Group #1 transgastric appendectomy:

1. Males and Females between the ages of 18-75
2. Clinical diagnosis of appendicitis Emergency room evaluation within 36 hours of the onset of pain
3. ASA classification I
4. Mentally competent to give informed consent.
5. Scheduled to undergo a transgastric NOTES appendectomy.

Exclusion criteria for group #1 transgastric appendectomy:

1. Pregnant women
2. Morbidly obese patients (Body mass index > 35)
3. Patients who are taking immunosuppressive medications or are immunocompromised
4. Patients who are on Proton Pump Inhibitors (PPI)
5. Patients with evidence of an abdominal abscess or mass on CT scan
6. Patients who present with a clinical diagnosis of sepsis
7. Patients who have a history of open abdominal surgery
8. Patients with diffuse peritonitis
9. Patients on blood thinners or aspirin

Inclusion criteria for Group #2 transgastric cholecystectomy:

1. Males and Females between the ages of 18 -75
2. Diagnosis of gallstone disease that require cholecystectomy
3. ASA classification I
4. Mentally competent to give informed consent.
5. Scheduled to undergo a transgastric NOTES cholecystectomy.

Exclusion criteria for Group #2 transgastric cholecystectomy:

1. Pregnant women
2. Patients with a Body mass index > 35
3. Patients who are taking immunosuppressive medications or are immunocompromised
4. Patients who are on Proton Pump Inhibitors (PPI)
5. Patients with suspicion of gallbladder cancer
6. Patients with a history of open abdominal surgery
7. Patients with known common bile duct stones (gallstones are not limited to the gallbladder)
8. Patients on blood thinners or aspirin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be 2 groups in this study: Of special note, the inclusion criteria clearly states subjects must be seen within 36 hours of the onset of pain and have an ASA Classification of I. This is intended to avoid obtaining informed consent from a subject who is in severe pain and incapable of making an informed decision, as well as avoid coercion. An ASA Classification of I defines a healthy normal individual.
  1. Group 1 will be transgastric laparoscopic assisted appendectomy
  2. Group 2 will be transgastric laparoscopic assisted cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2008-02; Primary Completion 2018-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of transgastric NOTES appendectomies and cholecystectomies (through data collection). | 1 year

SECONDARY OUTCOMES:
To evaluate pain associated with the transgastric approach (through data collection). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Horgan, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, San Diego, California, United States